CLINICAL TRIAL: NCT06313333
Title: Registro Nazionale Della Dermatite Atopica Moderata e Severa Nell'Adulto
Brief Title: National Register of Moderate and Severe Adult Atopic Dermatitis
Acronym: ATOPYREG
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana di Dermatologia Medica, Chirurgica, Estetica e di Malattie Sessualmente Trasmesse (Other)
Responsible Party: Sponsor
Other Study IDs: SID01
Record Dates: First submitted 2023-07-25; First posted 2024-03-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Collect clinical history and treatment data of AD in adulthood;

DETAILED DESCRIPTION:
Atopic dermatitis is a chronic-recurrent inflammatory skin disease with high prevalence in children and frequently presenting clinical remission during or after childhood; however, it may persist and/or recur, even after long and transient remission, adulthood. In addition, in some adult patients, DA is not present in pediatric age, but onset in adulthood: the investigators speak, in these cases, of adult-onset DA. The prevalence of DA is increasing all over the world and the cases in which clinical manifestations appear or persist during adolescence and/or adulthood are increased especially in industrialized countries. are not currently available specific laboratory markers for diagnosis of DA and, therefore, diagnosis is eminently clinical. In fact, at the present time, there are no validated diagnostic criteria, nor is there a clear consensus on diagnostic-therapeutic pathway to be followed when evaluating patients with adult DA. For these reasons, the collection of data related to various aspects of the DA such as those epidemiological, medical and clinical history, as well as the impact of the disease on the quality of life, results of crucial importance for estimating the real prevalence of this disease in Italy and also, possibly, to outline possible diagnostic criteria specific to adult DA, so that to facilitate and improve the diagnostic-therapeutic path of the patient. The intention of the project, therefore, is to create and use a National Register dedicated to DA patients in adulthood regardless of the period of onset of their pathology. aim to place the Italian Register as a supranational reference for international studies conducted on the adult DA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years
2. Signature of informed consent
3. Diagnosis of moderate and/or severe DA by a dermatologist specialist defined on the basis of following criteria (10):

   * EASI 16
   * EASI <16 but with at least one of the following conditions:

     1. location in at least one of the following "critical" locations: face, hands, genitals
     2. QID > 10
     3. VAS itching > 7
     4. VAS sleep > 7

Exclusion Criteria:

1. Patient unable to provide informed consent prior to any collection procedures data on the study;
2. unable to complete the procedures required for the study;
3. a patient already participating in another follow-up register of the same disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The nature of the study is descriptive. Each centre undertakes to recruit all adult patients diagnosed with moderate-severe atopic dermatitis observed at the center.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiological data | from baseline through study completion, an average of 3 year
  Reassessment of the epidemiology of AD
Identification of factors for specific treatment | from baseline through study completion, an average of 3 year
  Assessment of treatment profiles and identification of factors that determine the decision about the specific treatment of moderate and severe AD
clinical and therapeutic data | from baseline through study completion, an average of 3 year
  Assessment of any comorbidities;
characterization of diagnostic criteria | from baseline through study completion, an average of 3 year
  Outlining possible diagnostic criteria specific to AD in adults;
Assessment of possible conditioning factors | from baseline through study completion, an average of 3 year
  Evaluation of the natural history of AD and identification of possible conditioning factors;

CONTACTS AND LOCATIONS:
Overall Officials: Piergiacomo MD Calzavara Pinton, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided